CLINICAL TRIAL: NCT04293484
Title: Cortico-Spinal tDCS as Rehabilitative Intervention in Amyotrophic Lateral: a Randomized, Double-blind, Sham-controlled Trial Followed by an Open-label Phase
Brief Title: Cortico-Spinal tDCS as Rehabilitative Intervention in Amyotrophic Lateral Sclerosis
Acronym: tDCS_MND_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Prof., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP2743 v2
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Motor Neuron Disease, Familial; Amyotrophic Lateral Sclerosis With Dementia
Keywords: Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Transcranial direct current stimulation; tDCS; Non-invasive brain stimulation; Transcranial magnetic stimulation; TMS
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS - Real tDCS (Experimental): 10 sessions of anodal bilateral motor cortex and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks) followed by an open-label 10 sessions of anodal cerebellar and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Interventions: Device: Anodal bilateral motor cortex and cathodal spinal tDCS
- Sham tDCS - Real tDCS (Sham Comparator): 10 sessions of sham bilateral motor cortex and sham spinal transcranial direct current stimulation (5 days/week for 2 weeks) followed by an open-label 10 sessions of anodal cerebellar and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Interventions: Device: Anodal bilateral motor cortex and cathodal spinal tDCS; Device: Sham bilateral motor cortex and sham spinal tDCS

INTERVENTIONS:
Device: Anodal bilateral motor cortex and cathodal spinal tDCS — 10 sessions of anodal bilateral motor cortex and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks)
Device: Sham bilateral motor cortex and sham spinal tDCS — 10 sessions of sham bilateral motor cortex and sham spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Sham tDCS - Real tDCS

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a motor neuron disease, which is a group of neurological disorders that selectively affect motor neurons, the cells that control voluntary muscles of the body. The disorder causes muscle weakness and atrophy throughout the body due to the degeneration of the upper and lower motor neurons. Current drugs approved for ALS treatment only modestly slow disease progression.

Transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebral excitability in several neurodegenerative disorders and modulate intracortical connectivity measures.

In this randomized, double-blind, sham-controlled study followed by an open-label phase, the investigators will evaluate whether a repetition of two-weeks' treatment with bilateral motor cortex anodal tDCS and spinal cathodal tDCS, after a six months interval, may further outlast clinical improvement in patients with amyotrophic lateral sclerosis and can modulate intracortical connectivity, at short and long term.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a motor neuron disease, which is a group of neurological disorders that selectively affect motor neurons, the cells that control voluntary muscles of the body. The disorder causes muscle weakness and atrophy throughout the body due to the degeneration of the upper and lower motor neurons. Current drugs approved for ALS treatment only modestly slow disease progression.

Transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebral excitability in several neurodegenerative disorders and modulate intracortical connectivity measures.

The present randomized, double-blind, sham-controlled study followed by an open-label phase will investigate a repetition of two-weeks' treatment with bilateral motor cortex anodal tDCS and spinal cathodal tDCS, after a six months interval, may further outlast clinical improvement in patients with amyotrophic lateral sclerosis and modulate intracortical connectivity, at short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of probable, laboratory-supported probable, or definite amyotrophic lateral sclerosis according to the El Escorial revised criteria
* Disease duration ≤ 24 months
* Disease progression in the past 3 months
* Score ≥ 2 at the item "swallowing" of the ALS Functional Rating Scale Revised
* Score ≥ 2 at the item "walking" of the ALS Functional Rating Scale Revised
* Treatment with steady regimen of riluzole for a minimum of 1 month before study entry, and desiring its continuation
* Able to give informed consent
* Written informed consent

Exclusion Criteria:

* Motor neuron diseases other than ALS
* Severe head trauma in the past
* History of seizures
* History of ischemic stroke or hemorrhage
* Pacemaker
* Metal implants in the head/neck region
* Severe comorbidity
* Intake of illegal drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Strength From Baseline | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  A megascore is obtained by summing scores of single muscles (shoulder abductors, elbow flexors and extensors, wrist flexors, thumb opponent, hip flexors, knee flexors and extensors, and ankle dorsiflexors and extensors on both sides) manually evaluated according to the Medical Research Council (MRC) scale, which ranges from 0 (no movement) to 5 (normal contraction).
  The score for each muscle is summed, with scores ranging from 100 (no impairment) to 0 (most severe impairment).

SECONDARY OUTCOMES:
Change in Short-interval Intracortical Inhibition (SICI) From Baseline | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of tDCS on short-interval intracortical inhibition (SICI) from baseline
Change in the ALSFRS-R Score From Baseline | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  Change in the ALS Functional Rating Scale (ALSFRS-R) score from baseline. The ALSFRS provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. The ALSFRS includes ten questions that rate the patients level of functional impairment in performing one of ten common tasks. Each task is rated on a five-point scale from 0 (can't do) to 4 (normal ability). Individual item scores are summed to produce a reported score of between 40 (no impairment) and 0 (severe impairment).
Change of Quality of Life From Baseline: ALSAQ-40 Scale | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  Change of quality of life from baseline evaluated with the ALSAQ-40 scale. The Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ) is a patient self-report health status scale. The ALSAQ is specifically used to measure the subjective well-being of patients with amyotrophic lateral sclerosis. There are 40 items/questions with 5 discrete scales: physical mobility (10 items), activities of daily living and independence (10 items), eating and drinking (3 items), communication (7 items), emotional reactions (10 items). Patients are asked to think about the difficulties they may have experienced during the last two weeks (e.g. I have found it difficult to feed myself). Patients are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale):
  never/rarely/sometimes/often/always or cannot do at all. The total ranges from 0 (no impairment) to 160 (severe impairment).
Change of Quality of Life From Baseline: EQ-5D-5L Scale | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  Change of quality of life from baseline evaluated with the EQ-5D-5L scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The scale ranges from 5 (no impairment) to 25 (severe impairment).
Change of Quality of Life From Baseline: EQ-VAS Scale | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  Change of quality of life from baseline evaluated with the EQ-VAS scale. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. The scale ranges from 0 (severe impairment) to 100 (no impairment).
Change in Caregiver Burden (CBI) | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  Change of quality of life from baseline evaluated with the CBI scale. The CBI scale is 24- item scale designed to assess the experience of caregivers of older people. The multidimensional instrument assesses five domains of burden (time-dependence, developmental, physical, social, and emotional). Items are scored on a 4-point scale, ranging from "not at all descriptive" to "very descriptive". The scale ranges from 0 (no impairment) to 96 (severe impairment).
Change Intracortical Facilitation (ICF) From Baseline | Baseline - 2 weeks - 2 month - 6 months - 6 months and 2 weeks - 8 months - 12 months
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of tDCS on intracortical facilitation (ICF) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — Università degli Studi di Brescia; Alberto Benussi, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- AO Spedali Civili, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benussi A, Alberici A, Cotelli MS, Dell'Era V, Cantoni V, Bonetta E, Manenti R, Filosto M, Morini R, Datta A, Thomas C, Padovani A, Borroni B. Cortico-spinal tDCS in ALS: A randomized, double-blind, sham-controlled trial. Brain Stimul. 2019 Sep-Oct;12(5):1332-1334. doi: 10.1016/j.brs.2019.06.011. Epub 2019 Jun 8. No abstract available. PMID 31204206
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Menon P, Geevasinga N, Yiannikas C, Howells J, Kiernan MC, Vucic S. Sensitivity and specificity of threshold tracking transcranial magnetic stimulation for diagnosis of amyotrophic lateral sclerosis: a prospective study. Lancet Neurol. 2015 May;14(5):478-84. doi: 10.1016/S1474-4422(15)00014-9. Epub 2015 Apr 3. PMID 25843898
- [Background] Burrell JR, Kiernan MC, Vucic S, Hodges JR. Motor neuron dysfunction in frontotemporal dementia. Brain. 2011 Sep;134(Pt 9):2582-94. doi: 10.1093/brain/awr195. Epub 2011 Aug 11. PMID 21840887
- [Derived] Benussi A, Cantoni V, Grassi M, Libri I, Cotelli MS, Tarantino B, Datta A, Thomas C, Huber N, Karkkainen S, Herukka SK, Haapasalo A, Filosto M, Padovani A, Borroni B. Cortico-spinal tDCS in amyotrophic lateral sclerosis: A randomized, double-blind, sham-controlled trial followed by an open-label phase. Brain Stimul. 2023 Nov-Dec;16(6):1666-1676. doi: 10.1016/j.brs.2023.11.008. Epub 2023 Nov 15. PMID 37977335